CLINICAL TRIAL: NCT03922178
Title: Evaluation of Hemodynamic Changes of the Left Ventricle Following the Use of Extracorporeal Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Medical Director of the CHU Brugmann Hospital, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUB-Leclercq
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Coronary Surgery
MeSH Terms: interventions — Echocardiography; Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elective coronary surgery (Experimental): The study will be conducted at the CHU Brugmann Hospital, with collaboration between cardiac surgery and anesthesiology wards. Subjects referred for elective coronary surgery will be prospectively included during the length of the study.
  Interventions: Device: Pressure/Volume Combination Catheter; Device: Transthoracic echocardiography; Device: Transesophageal echocardiogram

INTERVENTIONS:
Device: Pressure/Volume Combination Catheter — Hemodynamic data routinely collected and data collected by means of the placement of a Pressure/Volume Combination Catheter (Pressure/Volume Combination Catheter,Leycom,The Netherlands) will be collected simultaneously. The catheter will be placed and held in place as long as the patient is in a position to be assisted by extracorporeal circulation. This means that the placement of the catheter will follow the heparinization of the patient and the placement of the cannulas necessary for the realization of extracorporal circulation. It will be removed from the left ventricular cavity before removal of extra-corporal cannulas.
Device: Transthoracic echocardiography — A complete transthoracic echocardiography will be performed the day before the surgical procedure, as per standard of care. It will establish the presence of the inclusion and exclusion criteria and evaluate the contractile function of the left ventricle. This will be done using a Philips IE33 echocardiograph (Koninklijke Philips Electronics N.V., Netherlands).
Device: Transesophageal echocardiogram — A transesophageal echocardiogram will be performed during the cardiac surgery, as per standard of care, using an Acuson Sequoia system (Siemens AG, Germany). It will facilitate the placement of the pressure/volume combination catheter and collect echographic data.

SUMMARY:
The interpretation of perioperative measures of cardiac function during cardiac surgery is complicated. In particular, the evaluation of the diastolic compliance of the left ventricle. In addition, they are subject to variations induced by post-charge changes caused by the anesthesia, extracorporeal circulation (ECC) and the surgical procedure itself.

Left ventricular failure is frequently measured by alteration of LV contractile properties, and very rarely by alteration of LV compliance. However, both contractility (systolic) and relaxation (diastolic) parameters are important for the left ventricle to perform its function adequately. Left ventricular failure after cardiac surgery with extracorporeal circulation and cardiac arrest under cardioplegia protection is an important and frequently reported complication. The investigator's objectives are to characterize the diastolic hemodynamic mechanisms of this left ventricular failure and to identify predictors of this failure in the postoperative period.

The quantification of the systolic and diastolic functions of the left ventricle by ventricular pressure-volume curves is the technique of reference today, because it allows to determine parameters that are independent of the pre- and post-load conditions. Previous studies using the conductance catheter for the purpose of estimating left ventricular function perioperatively are rare and report conflicting results. In addition, they were mainly intended to measure the systolic function of the left ventricle. Only one reported the diastolic relaxation parameters evaluated by a conductance catheter. This study showed immediately after withdrawal of the extracorporeal circulation a significant alteration of the diastolic relaxation of the left ventricle, but was not interested in its early (kinetic) evolution peroperatively.

The investigator's experience shows that, in the quarter-hour following the weaning of the extracorporeal circulation, a decrease in filling pressures of the left ventricle concomitant with an increase in cardiac output is objectified. These observations are consistent with a significant improvement in left ventricle compliance, but have never been reported.

The objectives of this study are:

* To characterize the left ventricular diastolic failure after withdrawal of the extracorporeal circulation in coronary surgery.
* To identify the kinetics of this early diastolic failure after withdrawal of the extracorporeal circulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the CHU Brugmann Hospital receiving elective coronary surgery.
* Patient in sinusal rhythm before the operation and during the collection of hemodynamic data.
* Patients with conserved left ventricular function (based on left ventricular ejection fraction assessed by preoperative echocardiography and superior to 50%)

Exclusion Criteria:

* Hypertrophic cardiomyopathy (diastolic septal thickness> 15 mm)
* Heart failure with left ventricular ejection fraction <50%
* Presence of cardiac valvulopathy, concerning both right and left atrio-ventricular and ventriculo-arterial valves
* Presence of valvular prosthesis
* Congenital heart disease
* Pregnancy
* Participation to another clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Tele-systolic pressure of the left ventricle | Baseline (before extracorporeal circulation is switched on)
  Pressure within the left ventricle after the atrial contraction, at the beginning of the ventricular contraction.
Tele-systolic pressure of the left ventricle | 1 minute after extracorporeal circulation is switched on
  Pressure within the left ventricle after the atrial contraction, at the beginning of the ventricular contraction.
Tele-systolic pressure of the left ventricle | 1 minute after extracorporeal circulation is stopped
  Pressure within the left ventricle after the atrial contraction, at the beginning of the ventricular contraction.
Tele-systolic pressure of the left ventricle | 10 minutes after extracorporeal circulation is stopped
  Pressure within the left ventricle after the atrial contraction, at the beginning of the ventricular contraction.
Tele-systolic pressure of the left ventricle | 20 minutes after extracorporeal circulation is stopped
  Pressure within the left ventricle after the atrial contraction, at the beginning of the ventricular contraction.
Diastolic pressure of the left ventricle | Baseline (before extracorporeal circulation is switched on)
  The pressure within the left ventricle following the completion of diastolic filling, just prior to systole.
Diastolic pressure of the left ventricle | 1 minute after extracorporeal circulation is switched on
  The pressure within the left ventricle following the completion of diastolic filling, just prior to systole.
Diastolic pressure of the left ventricle | 1 minute after extracorporeal circulation is stopped
  The pressure within the left ventricle following the completion of diastolic filling, just prior to systole.
Diastolic pressure of the left ventricle | 10 minutes after extracorporeal circulation is stopped
  The pressure within the left ventricle following the completion of diastolic filling, just prior to systole.
Diastolic pressure of the left ventricle | 20 minutes after extracorporeal circulation is stopped
  The pressure within the left ventricle following the completion of diastolic filling, just prior to systole.
Tele-systolic volume of the left ventricle | Baseline
  At the end of systole, the ventricle contains a quantity of blood called 'telesystolic volume'.
Tele-systolic volume of the left ventricle | 1 minute after extracorporeal circulation is switched on
  At the end of systole, the ventricle contains a quantity of blood called 'telesystolic volume'.
Tele-systolic volume of the left ventricle | 1 minute after extracorporeal circulation is stopped
  At the end of systole, the ventricle contains a quantity of blood called 'telesystolic volume'.
Tele-systolic volume of the left ventricle | 10 minutes after extracorporeal circulation is stopped
  At the end of systole, the ventricle contains a quantity of blood called 'telesystolic volume'.
Tele-systolic volume of the left ventricle | 20 minutes after extracorporeal circulation is stopped
  At the end of systole, the ventricle contains a quantity of blood called 'telesystolic volume'.
Diastolic volume of the left ventricle | Baseline
  At the end of diastole, the ventricle contains a quantity of blood called end-diastolic volume.
Diastolic volume of the left ventricle | 1 minute after extracorporeal circulation is switched on
  At the end of diastole, the ventricle contains a quantity of blood called end-diastolic volume.
Diastolic volume of the left ventricle | 1 minute after extracorporeal circulation is stopped
  At the end of diastole, the ventricle contains a quantity of blood called end-diastolic volume.
Diastolic volume of the left ventricle | 10 minutes after extracorporeal circulation is stopped
  At the end of diastole, the ventricle contains a quantity of blood called end-diastolic volume.
Diastolic volume of the left ventricle | 20 minutes after extracorporeal circulation is stopped
  At the end of diastole, the ventricle contains a quantity of blood called end-diastolic volume.
Ejection volume of the left ventricle | Baseline
  The ejection volume is the difference between systolic and diastolic volume. It represents the amount of blood ejected at each contraction by the ventricle.
Ejection volume of the left ventricle | 1 minute after extracorporeal circulation is switched on
  The ejection volume is the difference between systolic and diastolic volume. It represents the amount of blood ejected at each contraction by the ventricle.
Ejection volume of the left ventricle | 1 minute after extracorporeal circulation is stopped
  The ejection volume is the difference between systolic and diastolic volume. It represents the amount of blood ejected at each contraction by the ventricle.
Ejection volume of the left ventricle | 10 minutes after extracorporeal circulation is stopped
  The ejection volume is the difference between systolic and diastolic volume. It represents the amount of blood ejected at each contraction by the ventricle.
Ejection volume of the left ventricle | 20 minutes after extracorporeal circulation is stopped
  The ejection volume is the difference between systolic and diastolic volume. It represents the amount of blood ejected at each contraction by the ventricle.
Contractility index of the left ventricle | Baseline
  Computed by the following formula: (dP/dt max)/P
Contractility index of the left ventricle | 1 minute after extracorporeal circulation is switched on
  Computed by the following formula: (dP/dt max)/P
Contractility index of the left ventricle | 1 minute after extracorporeal circulation is stopped
  Computed by the following formula: (dP/dt max)/P
Contractility index of the left ventricle | 10 minutes after extracorporeal circulation is stopped
  Computed by the following formula: (dP/dt max)/P
Contractility index of the left ventricle | 20 minutes after extracorporeal circulation is stopped
  Computed by the following formula: (dP/dt max)/P

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Leclercq, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No